CLINICAL TRIAL: NCT01788891
Title: TASER-Pediatrics: Prospective Monitoring of Second-line Antiretroviral Therapy Failure and Resistance in Children
Brief Title: Second-line Therapy
Acronym: TASER-P
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other); Dr Cipto Mangunkusumo General Hospital (Other); Pediatric Institute, Hospital Kuala Lumpur (Unknown); Chiang Mai University (Other); Srinagarind Hospital, Khon Kaen University (Other); Mahidol University (Other); Children's Hospital Number 1, Ho Chi Minh City, Vietnam (Other); Number 2 Children's Hospital, Ho Chi Minh City (Other); Kirby Institute (Other Government); University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 149
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Treatment Failure of Second-line ART in Asian HIV-infected Children
Keywords: longitudinal observational cohort study; multicenter; pediatrics; Asian; treatment failure; renal status; toxicities; therapeutic drug monitoring (TDM); drug levels in blood and hair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and hair will be used for therapeutic drug monitoring (TDM). Blood drawn at every visit will be used to assess CD4 count, viral load, and other basic chemistry test panel. If necessary, drug resistant tests will also be carried out on the blood samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- second-line pediatric cohort: Asian HIV-positive children <18 years old who are receiving HIV care at one of the participating TREAT Asia Pediatric HIV Observational Database (TApHOD) sites that have been identified for TASER-P participation will be monitored for treatment failure of second-line ART

SUMMARY:
This study will help identify which ARV candidates should be prioritized for pediatric use in resource-limited settings

DETAILED DESCRIPTION:
Children in resource-limited settings are increasing experiencing treatment failure, as defined by virologic, immunologic, and/or clinical criteria. There are few studies of HIV resistance mutations in children failing first line NNRTI therapy in resource limited settings. The emergence of treatment failure and drug resistance in children on ART emphasizes the urgency for developing evidence-based second-line and salvage treatment strategies. Pediatric treatment is complicated by a number of factors, including having fewer numbers of ARVs approved by drug safety agencies and the lack of pediatric formulations. This further shortens the list of available second-line ARVs as compared to adults.

Despite the growing number of children on second-line therapy worldwide, there are limited data on efficacy of second-line PI therapy in children after NRTI-NNRTI failure. There are currently no options for third-line/salvage regimens for children in resource-limited settings. New drugs and drug classes are approved for use in children by the US FDA but are not routinely available outside of high-income settings.

Also, there are no data on the resistance patterns of children failing second-line therapy in resource-limited settings to guide clinical management and ARV procurement. Clinicians need evidence-based guidelines for how to manage children with treatment failure, and access to the drugs necessary to construct potent and durable third-line regimens.

TASER-P is a longitudinal observational cohort study to monitor for treatment failure to second-line ART in Asian children.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years old
* Have confirmed HIV infection
* Are being switched to or treated with second-line ART. Second-line ART is defined as the second regimen with a major antiretroviral class switch. For example, a switch from an NNRTI-based to a PI-based regimen or vice versa
* Caregivers give informed consent. Children will be asked to give assent if they know their HIV status and have reached the minimum age to give assent according to each site's institutional review board regulations

Exclusion Criteria:

* Started mono- or dual- therapy as the first ART therapy
* Failing first-line triple nucleoside reverse transcriptase inhibitor regimen
* Are being switched to or treated with second-line ART without failure of first-line therapy (i.e., for toxicity)
* Caregiver +/- child (if asked to give assent) refuses to participate in this study
* Have not been enrolled in TApHOD

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HIV-positive children <18 years old who are have switched to or treated with second-line ART at one of the participating TREAT Asia Pediatric HIV Observational Database (TApHOD) sites.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
resistance | week 72
  To monitor for resistance development and resistance patterns in children failing second-line ART over 72 weeks

SECONDARY OUTCOMES:
virologic failure | week 72
  To determine the frequency of virologic suppression defined as HIV-RNA <400 copies/ml over 72 weeks To determine the frequency of virologic failure as HIV RNA ≥1000 copies/ml over 72 weeks To evaluate predictors of virologic failure
drug resistance | week 72
  To assess HIV drug resistance patterns by virtual phenotyping
ARV drug levels | week 72
  To correlate ARV drug levels between plasma and hair samples To correlate hair ARV levels with virologic responses and measures of adherence

CONTACTS AND LOCATIONS:
Overall Officials: Nia Kurniati, MD, Principal Investigator — Dr Cipto Mangunkusumo General Hospital; Kamarul Razali, MD, Principal Investigator — Kuala Lumpur General Hospital; Tavitiya Sudjaritruk, MD, Principal Investigator — Research Institute for Health Sciences, Chiang Mai University; Pope Kosalaraksa, MD, Principal Investigator — Srinagarind Hospital, Khon Kaen Hospital; Kulkanya Chokephaibulkit, MD, Principal Investigator — Siriraj Hospital; Truong Huu Khanh, MD, Principal Investigator — Children's Hospital Number 1; Do Chau Viet, MD, Principal Investigator — Children's Hospital Number 2; Jintanat Ananworanich, MD, PhD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration; Annette Sohn, MD, Principal Investigator — TREAT Asia
Locations (8):
- Mangunkusumo General Hospital, Jakarta, Indonesia
- Hospital Kuala Lumpur, Kuala Lumpur, Malaysia
- Thailand (4):
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen, Changwat Khon Kaen
  - Research Institute for Health Sciences, Chiang Mai, Chiang Mai
  - HIV-NAT, Bangkok
  - Siriraj Hospital, Bangkok
- Vietnam (2):
  - Children's Hospital Number 1, Ho Chi Minh City
  - Children's Hospital Number 2, Ho Chi Minh City

REFERENCES:
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT)'s website — http://www.hivnat.org